CLINICAL TRIAL: NCT01316874
Title: Intravesical AD 32 (Valrubicin) in Patients With Carcinoma in Situ (CIS) of the Bladder Who Have Failed or Have Recurrence Following Treatment With Bacillus Calmette-Guerin (BCG)
Acronym: Bladder Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director Clinical R&D, Endo Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9301/A9302
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Carcinoma in Situ; Bladder Cancer
Keywords: Valrubicin; CIS; AD 32, BCG-refractory CIS; Carcinoma in situ (CIS) previously treated with BCG
MeSH Terms: conditions — Carcinoma in Situ; Urinary Bladder Neoplasms | interventions — valrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AD32 (valrubicin) (Experimental): 800mg, once weekly for 6 weeks
  Interventions: Drug: Valrubicin, 800 mg

INTERVENTIONS:
Drug: Valrubicin, 800 mg — Investigator will be responsible for regulating the use of concomitant medications (systemic and/or topical anticholinergic therapy or topical anesthesia) and other medications.

SUMMARY:
This is a Phase II/Phase III study of intravesical AD 32 (valrubicin) in patients with carcinoma in situ (CIS) who have been previously treated with intravesical Bacillus Calmette-Guerin (BCG) for CIS and in whom recurrence or failure has occurred after multiple courses of intravesical treatment.

ELIGIBILITY:
Inclusion-

1. Patients must have pathologically-proven CIS with no evidence of muscle invasive disease.
2. Patients with concurrent Ta or T1 papillary tumors are eligible provided papillary tumor(s) are resected prior to study treatment. Cystoscopic evaluation and, if indicated, transurethral resection of bladder tumor (TURBT) must be performed within 28 days of study treatment.
3. Patients must have received at least two or more prior courses of intravesical therapy for CIS per the recommended schedules. BCG must have been one of the prior therapies administered. Patients can have either failed BCG therapy or have been successfully treated with BCG, but subsequently found to have recurrence. The standard course of intravesical therapy must include six weekly treatments (allowable range of instillations per course is 4-9).
4. Patients must have a positive urine cytology at baseline (<28 days) prior to the first AD 32 (valrubicin) treatment. Patients with papillary lesions must have a positive cytology following TURBT or have a baseline cytology that was negative or equivocal and histologic confirmation of CIS.
5. Patients must have an ECOG performance status of 0-2 and a life expectancy of at least 6 months.

Exclusion-

1. Patients with urogenital tumors with histology other than transitional cell carcinoma
2. Patients with residual papillary disease at the time of study treatment.
3. Patients with a history of other primary malignancy (other than squamous or basal cell skin cancers) within the last 5 years.
4. Patients with evidence of muscle invasive disease (stage higher than T1).
5. Patients with any previous intravesical treatment with AD 32 (valrubicin).
6. Patients with any intravesical therapy within 28 days prior to first AD 32 (valrubicin) treatment.
7. Patients with a plan to receive other concurrent therapy for treatment of primary treatment tumor during participation in this study.
8. Patients who had received prior systemic or radiation therapy for bladder cancer.
9. Women who were pregnant or lactating. Individuals of reproductive potential could not participate unless agreeing to use an effective contraceptive method for themselves and/or their sexual partners.
10. Patients who, in the investigator's opinion, could not comply with the provisions of the protocol or did not understand the nature of the study.
11. Patients who, in the opinion of the investigator, could not tolerate intravesical administration of approximately 75 mL of fluid or who could not tolerate surgical manipulation (cystoscopy, mapping biopsies, barbotage) due to the presence of concomitant serious illnesses (ie, uncontrolled cardiac or respiratory disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 1993-11; Primary Completion 1997-04 (Actual); Study Completion 1997-04 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of AD 32 (valrubicin) in patients with CIS of the bladder who previously have been treated with BCG for CIS and in whom recurrence or failure had occurred after multiple courses of intravesical treatment. | 12 weeks

SECONDARY OUTCOMES:
To evaluate the qualitative toxicities associated with intravesical therapy using AD 32 (valrubicin). | 6 weeks
To determine the concentration of anthracyclines in the voided urine of patients who chose to participate in a urine recovery study. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Stacy Childs, MD, Alabaster, Alabama
  - William Bohnert, MD, Phoenix, Arizona
  - Scott Swanson, MD, Scottsdale, Arizona
  - Bruce Dalkin, MD, Tucson, Arizona
  - Donald Gleason, MD, Tucson, Arizona
  - William Friedel, MD, La Mesa, California
  - Stephen Auerbach, MD, Newport Beach, California
  - William Moseley, MD, San Diego, California
  - Standley Brosman, MD, Santa Monica, California
  - Eugene Dula, MD, Van Nuys, California
  - B. Thomas Brown, MD, Daytona Beach, Florida
  - Charles Jackson, MD, Fort Lauderdale, Florida
  - Marc Soloway, MD, Miami, Florida
  - Charles Brendler, MD, Chicago, Illinois
  - Patrick Guinan, MD, Chicago, Illinois
  - Jeffrey Ignatoff, MD, Evanston, Illinois
  - David Wood, MD, Lexington, Kentucky
  - John Tuttle, MD, Lexington, Kentucky
  - Dennis Venable, MD, Shreveport, Louisiana
  - Harold Frazier, MD, Bethasda, Maryland
  - Myron Murdock, MD, Greenbelt, Maryland
  - John Libertino, Burlington, Massachusetts
  - W. Lamar Weems, MD, Jackson, Mississippi
  - Hugh Fisher, MD, Albany, New York
  - Michael Blute, MD, Rochester, New York
  - Michael Wolff, MD, Burlington, North Carolina
  - Cary Robertson, MD, Durham, North Carolina
  - Eric Klein, MD, Cleveland, Ohio
  - Bruce Lowe, MD, Portland, Oregon
  - Jeffrey Cohen, MD, Pittsburgh, Pennsylvania
  - Jacques Susset, MD, Providence, Rhode Island
  - L. Dean Knoll, MD, Nashville, Tennessee
  - Steohen Hardeman, MD, Austin, Texas
  - Ian Thompson, MD, Fort San Houston, Texas
  - Seth Lemer, MD, Houston, Texas
  - Aaron Katz, MD, Richmond, Virginia
  - Gary Katz, MD, Richmond, Virginia
  - Williams Ellis, MD, Seattle, Washington
  - Richard Boxer, MD, Milwaukee, Wisconsin

REFERENCES:
- [Background] Steinberg G, Bahnson R, Brosman S, Middleton R, Wajsman Z, Wehle M. Efficacy and safety of valrubicin for the treatment of Bacillus Calmette-Guerin refractory carcinoma in situ of the bladder. The Valrubicin Study Group. J Urol. 2000 Mar;163(3):761-7. PMID 10687972
- [Derived] Steinberg GD, Smith ND, Ryder K, Strangman NM, Slater SJ. Factors affecting valrubicin response in patients with bacillus Calmette-Guerin-refractory bladder carcinoma in situ. Postgrad Med. 2011 May;123(3):28-34. doi: 10.3810/pgm.2011.05.2281. PMID 21566413